CLINICAL TRIAL: NCT04560530
Title: The Use of Preoperative CT Chest Scan in the Pre-anesthetic Assessment of COVID-19
Brief Title: The Role of CT Chest Scan in the Pre-anesthetic Assessment of Suspected or Confirmed COVID -19 Patients
Status: Completed | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, MOHAMMED FAWZI ALI ABOSAMAK, ICU consultant, Tanta University
Other Study IDs: chest CT scan in COVID-19
Record Dates: First submitted 2020-09-22; First posted 2020-09-23 (Actual); Last update posted 2020-09-23 (Actual); Status verified 2020-09

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Non-enhanced CT scan of the chest — Non-enhanced CT scan of the chest with multi-slice CT scan machine.

SUMMARY:
The role of CT scan of the chest in Pre-anesthetic assessment of the severity of COVID-19 and the correlations between CT measurements of the aortic and pulmonary arteries diameters and severity of pneumonia.

DETAILED DESCRIPTION:
Patients who were scheduled for emergency surgery during COVID-19 pandemic should have be screened for COVID pre-operatively given the prevalence f asymptomatic or mildly symptomatic cases that could be carriers to infection and possibly cause cross infection to the operating room staff especially the anesthetists who deal with the upper airway during intubation with high possibility of getting infected with SARS-COV 2 virus. Waiting respiratory tract PCR (RT-PCR) test for COVID can delay the surgery which may increase patients morbidity and mortality. RT-PCR test has limited sensitivity and specificity.

Patients who are confirmed to have COVID-19 infection (have positive RT-PCR) or patients who have possible COVID-19 infection (have symptoms but were not tested with RT-PCR) will undergo non-enhanced CT scanning of the chest (without giving IV contrast).

Chest CT scan will be interpreted by 2 Consultants radiologists with an experience of at least 10 years in their field.

The radiologists are going to be requested to comment on the lung parenchyma, describing the findings , assess the pulmonary artery, aorta diameters and the aorta:pulmonary diameters ratio will be then calculated. The degree of pneumonia severity index will then be described as well.

The radiologists will be blinded to the aim of the study.

All data will be collected and then correlation between the data sets will be statistically tested.

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for emergency surgery with symptoms suggestive of COVID-19 infection.

Exclusion Criteria:

* Pregnancy.
* Haemodynamic instability (Mean arterial blood pressure above 65 mmHg or the need for of inotropic drugs to maintain mean arterial blood pressure above 65 mmHg).
* Active bleeding.
* Any indication by the surgeon or the anesthesiologist to proceed for immediate surgery for the patient safety.
* Patients refusal to do CT scanning.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who are older than 18 years, having confirmed or suspected COVID-19 infection and scheduled for emergency surgery.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
pneumonia severity. | 90 days
  The pneumonia severity will be assessed by the radiologist.
Aorta diameter | 90 days
  Aorta cross sectional diameter will be calculated by using cursor method on CT scan
Pulmonary artery diameter | 90 days
  Pulmonary artery sectional diameter will be calculated by using cursor method on CT scan
Pulmonary artery diameter TO Aorta diameter ratio | 90 days
  Pulmonary artery diameter TO Aorta diameter ratio will be calculated

SECONDARY OUTCOMES:
Description of the lesions found in the CT scan | 90 days
  The parenchymal lesions will be described by the radiologist

CONTACTS AND LOCATIONS:
Locations (1):
- Security Forces Hospital, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided